CLINICAL TRIAL: NCT04784533
Title: A Study to Evaluate Maintenance of Hair Regrowth Following Dose Reduction of CTP-543 in Adult Patients With Moderate to Severe Alopecia Areata
Brief Title: A Study to Evaluate the Durability of Response of CTP-543 in Adult Patients With Moderate to Severe Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP543.2004
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Alopecia Areata
Keywords: CTP-543
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Part A: Period 1 - CTP-543 8 mg BID (Experimental): Participants received CTP-543 8 milligrams (mg) tablets, orally, twice daily (BID) for up to 24 weeks.
  Interventions: Drug: CTP-543
- Part A: Period 1 - CTP-543 12 mg BID (Experimental): Participants received CTP-543 12 mg tablets, orally, BID for up to 24 weeks.
  Interventions: Drug: CTP-543
- Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID (Experimental): Participants who received CTP-543 8 mg during Period 1 of Part A and achieved an absolute severity of alopecia tool (SALT) score of ≤20 at Week 24, received CTP-543 4 mg tablets, orally, BID, for up to 24 weeks.
  Interventions: Drug: CTP-543
- Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID (Experimental): Participants who received CTP-543 12 mg during Period 1 of Part A and achieved an absolute SALT score of ≤20 at Week 24, received CTP-543 8 mg tablets, orally, BID, for up to 24 weeks.
  Interventions: Drug: CTP-543
- Part A: Period 2 - CTP-543 8 mg BID to Placebo (Placebo Comparator): Participants who received CTP-543 8 mg during Period 1 of Part A and achieved an absolute SALT score of ≤20 at Week 24, received CTP-543 matched placebo tablets, orally, BID, for up to 24 weeks.
  Interventions: Drug: Placebo
- Part A: Period 2 - CTP-543 12 mg BID to Placebo (Placebo Comparator): Participants who received CTP-543 12 mg during Period 1 of Part A and achieved an absolute SALT score of ≤20 at Week 24, received CTP-543 matched placebo tablets, orally, BID, for up to 24 weeks.
  Interventions: Drug: Placebo
- Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID (Experimental): Participants who received CTP-543 8 mg during Period 1, followed by CTP-543 4 mg during Period 2 of Part A and met the criteria for loss of regrowth maintenance (LOM) (absolute SALT score of > 20), received re-treatment with CTP-543 8 mg tablets, orally, BID, for up to 24 weeks.
  Interventions: Drug: CTP-543
- Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID (Experimental): Participants who received CTP-543 12 mg during Period 1, followed by CTP-543 8 mg during Period 2 of Part A and met the criteria for LOM (absolute SALT score of > 20), received re-treatment with CTP-543 12 mg tablets, orally, BID, for up to 24 weeks.
  Interventions: Drug: CTP-543
- Part B: CTP-543 8 mg BID to Placebo to 8 mg BID (Experimental): Participants who received CTP-543 8 mg during Period 1, followed by CTP-543 matched placebo during Period 2 of Part A and met the criteria for LOM (absolute SALT score of > 20), received re-treatment with CTP-543 8 mg tablets, orally, BID, for up to 24 weeks.
  Interventions: Drug: CTP-543
- Part B: CTP-543 12 mg BID to Placebo to 12 mg BID (Experimental): Participants who received CTP-543 12 mg during Period 1, followed by CTP-543 matched placebo during Period 2 of Part A and met the criteria for LOM (absolute SALT score of > 20), received re-treatment with CTP-543 12 mg tablets, orally, BID, for up to 24 weeks.
  Interventions: Drug: CTP-543

INTERVENTIONS:
Drug: CTP-543 — Oral dosing
  Arms: Part A: Period 1 - CTP-543 12 mg BID; Part A: Period 1 - CTP-543 8 mg BID; Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID; Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID; Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID; Part B: CTP-543 12 mg BID to Placebo to 12 mg BID; Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID; Part B: CTP-543 8 mg BID to Placebo to 8 mg BID
Drug: Placebo — Oral dosing
  Arms: Part A: Period 2 - CTP-543 12 mg BID to Placebo; Part A: Period 2 - CTP-543 8 mg BID to Placebo

SUMMARY:
This study is designed to evaluate the regrowth of hair with CTP-543 and subsequent durability of that regrowth following dose reduction in adult patients with moderate to severe alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of alopecia areata with a current episode of scalp hair loss lasting at least 6 months and not exceeding 10 years at the time of Screening. Total disease duration greater than 10 years is permitted.
* At least 50% scalp hair loss, as defined by a severity of alopecia tool (SALT) score ≥50, at Screening and Baseline.
* Willing to comply with the study visits and requirements of the study protocol.

Exclusion Criteria:

* Treatment with other medications or agents within 1 month of Baseline or during the study that may affect hair regrowth or immune response.
* Active scalp inflammation, psoriasis, or seborrheic dermatitis requiring topical treatment to the scalp, significant trauma to the scalp, or other scalp condition that may interfere with the SALT assessment, or untreated actinic keratosis anywhere on the body at Screening and/or Baseline.
* Treatment with systemic immunosuppressive medications within 3 months of Screening or during the study, or biologics within 6 months of Screening or during the study.
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study drug.
* Clinically significant medical condition, psychiatric disease, or social condition, as determined by the Investigator, that may unfavorably alter the risk-benefit of study participation, adversely affect study compliance, or confound interpretation of study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Center for Dermatology and Plastic Surgery/CCT Research, Scottsdale, Arizona
  - Kern Research, Inc., Bakersfield, California
  - Hope Clinical Research, Canoga Park, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - University of California, Irvine, Irvine, California
  - Quest Dermatology Research, Northridge, California
  - Kaiser Permanente, Oakland, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - Kaiser Permanente, San Francisco, California
  - Colorado Center for Dermatology and Skin Surgery, Centennial, Colorado
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - Yale University Church Street Research Unit, New Haven, Connecticut
  - Skin Care Research, LLC, Boca Raton, Florida
  - Skin Care Research, LLC, Hollywood, Florida
  - DeNova Research, Chicago, Illinois
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - DS Research, Louisville, Kentucky
  - Michigan Center for Research Company, LLC, Clarkston, Michigan
  - University of Minnesota Department of Dermatology, Minneapolis, Minnesota
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - Skin Laser and Surgery Specialists of New Jersey, Hackensack, New Jersey
  - Darst Dermatology, Charlotte, North Carolina
  - Dermatology Specialists of Charlotte, Charlotte, North Carolina
  - North Carolina Dermatology Associates, PLLC, Raleigh, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Remington Davis, Columbus, Ohio
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Northwest Dermatology, Portland, Oregon
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - PEAK Research, LLC, Upper Saint Clair, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Dermatology Treatment and Research Center, PA, Dallas, Texas
  - Austin Institute for Clinical Research, Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Springville Dermatology/CCT Research, Springville, Utah
  - West End Dermatology Associates, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in the United States from 26 February 2021 to 16 May 2023.
Pre-assignment Details: 429 participants were screened, out of which 317 participants who experienced moderate to severe hair loss due to alopecia areata were enrolled to receive CTP-543 or placebo.
Period: Part A: Period 1 (Day 1 to Week 24)
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID | Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID | Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID | Part A: Period 2 - CTP-543 8 mg BID to Placebo | Part A: Period 2 - CTP-543 12 mg BID to Placebo | Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID
Started | 180 | 137 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Efficacy Population (Efficacy population included all participants who were randomized in the study, dispensed study drug, and had at least 1 post treatment severity of alopecia tool (SALT) assessment.) | 178 | 135 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 162 | 118 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 18 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment Emergent or Worsening Adverse Event | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance With Study Drug | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 5 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Period 2 (Week 24 to Week 48)
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID | Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID | Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID | Part A: Period 2 - CTP-543 8 mg BID to Placebo | Part A: Period 2 - CTP-543 12 mg BID to Placebo | Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID
Started (The Part A Period 2 consists of participants from Part A Period 1 from each dose group who achieved an absolute SALT score of ≤20 at Week 24.) | 0 | 0 | 18 | 25 | 18 | 25 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 17 | 25 | 18 | 25 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Day 1 to Week 24)
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID | Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID | Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID | Part A: Period 2 - CTP-543 8 mg BID to Placebo | Part A: Period 2 - CTP-543 12 mg BID to Placebo | Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID
Started (The Part B consists of participants who achieved loss of regrowth maintenance (absolute SALT score of > 20) from Part A Period 2.) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 15 | 19
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 13 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants included all participants who were randomized in the study.
Groups:
- Part A: Period 1 - CTP-543 8 mg BID: Participants received CTP-543 8 mg tablets, orally, BID for up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID | Total
Number analyzed (Participants) | 180 | 137 | 317
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (14.05) | 39.6 (13.21) | 39.8 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 93 | 212
  Male | 61 | 44 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 24
  Not Hispanic or Latino | 167 | 126 | 293
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 14 | 9 | 23
  Race: Black or African American | 41 | 24 | 65
  Race: Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Race: White | 121 | 102 | 223
  Race: Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part A, Period 2: Percentage of Participants Achieving Loss of Regrowth Maintenance (LOM) Criteria Defined by Severity of Alopecia Tool (SALT) Score > 20 Following Dose Reduction
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss). LOM is defined as an absolute SALT score >20. The percentage of participants achieving LOM criteria (SALT >20) was compared to the percentage of participants maintaining treatment success (SALT ≤ 20) for each of the following dose reduction conditions. Due to the variable time on study for each participant within Part A Period 2, the primary analysis visit was the end of Part A Period 2, where the last observed non-missing SALT value was selected for each participant.
Time Frame: From Week 24 to Week 48
Population: Efficacy Population included all participants who were randomized, dispensed study drug, and had at least 1 post-treatment SALT assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID: Participants who received CTP-543 8 mg during Period 1 of Part A and achieved an absolute SALT score of ≤20 at Week 24, received CTP-543 4 mg tablets, orally, BID, for up to 24 weeks.
Arm/Group | Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID | Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID
Number analyzed (Participants) | 18 | 25
Percentage of participants | 27.8 [7.1 to 48.5] | 32.0 [13.7 to 50.3]

2. Primary Outcome: Part A, Period 2: Percentage of Participants Achieving LOM Criteria Defined by SALT Score > 20 Following Drug Discontinuation
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss). LOM is defined as an absolute SALT score >20. The percentage of participants achieving LOM criteria (SALT >20) was compared to the percentage of participants maintaining treatment success (SALT ≤ 20) for each of the following dose discontinuation conditions. Due to the variable time on study for each participant within Part A Period 2, the primary analysis visit was at the end of Part A Period 2, where the last observed non-missing SALT value was selected for each participant.
Time Frame: From Week 24 to Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part A: Period 2 - CTP-543 8 mg BID to Placebo: Participants who received CTP-543 8 mg during Period 1 of Part A and achieved an absolute SALT score of ≤20 at Week 24, received CTP-543 4 mg tablets, orally, BID, for up to 24 weeks.
- Part A: Period 2 - CTP-543 12 mg BID to Placebo: Participants who received CTP-543 12 mg during Period 1 of Part A and achieved an absolute SALT score of ≤20 at Week 24, received CTP-543 8 mg tablets, orally, BID, for up to 24 weeks.
Arm/Group | Part A: Period 2 - CTP-543 8 mg BID to Placebo | Part A: Period 2 - CTP-543 12 mg BID to Placebo
Number analyzed (Participants) | 18 | 25
Percentage of participants | 83.3 [66.1 to 100.0] | 80.0 [64.3 to 95.7]

3. Primary Outcome: Part B: Percentage of Participants by Dose Group Who Achieved Restoration of Regrowth (ROR) at Week 24
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss). ROR is defined as the participant's attainment of an absolute SALT score of ≤20 at Week 24 of re-treatment.
Time Frame: Week 24 of re-treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID
Number analyzed (Participants) | 5 | 8 | 15 | 19
Percentage of participants | 60.0 [17.1 to 100.0] | 50.0 [15.4 to 84.6] | 66.7 [54.0 to 99.8] | 73.7 [58.6 to 97.0]

4. Secondary Outcome: Part A, Period 2: Percentage of Participants Who Achieved LOM Criteria Defined by SALT Score > 20 Following Dose Reduction Conditions at Weeks 28, 32, 36, 40, 44, and 48
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss). LOM is defined as an absolute SALT score >20.
Time Frame: Weeks 28, 32, 36, 40, 44, and 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID | Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID
Number analyzed (Participants) | 18 | 25
Percentage of participants
  Week 28 | 0 [NA to NA] — Not estimable as 0 participants achieved LOM criteria of SALT Score > 20 | 12 [2.5 to 31.2]
  Week 32 | 6.3 [0.2 to 30.2] | 4.5 [0.1 to 22.8]
  Week 36 | 0 [NA to NA] — Not estimable as 0 participants achieved LOM criteria of SALT Score > 20 | 4.8 [0.1 to 23.8]
  Week 40 | 12.5 [1.6 to 38.3] | 10.5 [1.3 to 33.1]
  Week 44 | 7.7 [0.2 to 36.0] | 0 [NA to NA] — Not estimable as 0 participants achieved LOM criteria of SALT Score > 20
  Week 48 | 7.7 [0.2 to 36.0] | 5.6 [0.1 to 27.3]

5. Secondary Outcome: Part A, Period 2: Percentage of Participants Who Achieved LOM Criteria Defined by SALT > 20 Following Drug Discontinuation Conditions at Weeks 28, 32, 36, 40, 44, and 48
Description: as for outcome 4
Time Frame: Weeks 28, 32, 36, 40, 44, and 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part A: Period 2 - CTP-543 8 mg to Placebo: Participants who responded with an absolute SALT score of ≤20 at week 24 of the treatment period with 8 mg in Period 1, received CTP-543-matched placebo tablets, orally, for up to 24 weeks.
- Part A, Period 2 - CTP-543 12 mg to CTP-543 Matched Placebo: Participants who responded with an absolute SALT score of ≤20 at week 24 of the treatment period with 12 mg in Period 1, received CTP-543 matched placebo tablets, orally, for up to 24 weeks
Arm/Group | Part A: Period 2 - CTP-543 8 mg to Placebo | Part A, Period 2 - CTP-543 12 mg to CTP-543 Matched Placebo
Number analyzed (Participants) | 18 | 25
Percentage of participants
  Week 28 | 0 [NA to NA] — Not estimable as 0 participants achieved LOM criteria of SALT Score > 20 | 16.7 [4.7 to 37.4]
  Week 32 | 16.7 [3.6 to 41.4] | 14.3 [3.0 to 36.3]
  Week 36 | 26.7 [7.8 to 55.1] | 43.8 [19.8 to 70.1]
  Week 40 | 36.4 [10.9 to 69.2] | 22.2 [2.8 to 60.0]
  Week 44 | 28.6 [3.7 to 71.0] | 0 [NA to NA] — Not estimable as 0 participants achieved LOM criteria of SALT Score > 20
  Week 48 | 40.0 [5.3 to 85.3] | 28.6 [3.7 to 71.0]

6. Secondary Outcome: Part A, Period 1: Percentage of Responders as Assessed on the Hair Satisfaction Patient Reported Outcome (SPRO) Scale at Weeks 12, 16, 20, and 24
Description: SPRO is a questionnaire answered by the participant and designed to measure how satisfied alopecia areata participants are with their hair at the time of the assessment. The responses range from 1 to 5: 1= very satisfied, 2= satisfied, 3= neither satisfied nor dissatisfied, 4= dissatisfied, and 5= very dissatisfied. SPRO responder is defined as a post-baseline response of 'very satisfied' or 'satisfied'.
Time Frame: Weeks 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part A: Period 1 - CTP-543 8 mg BID: Participants received CTP-543 8 mg tablets, orally, BID, for up to 24 weeks.
- Part A: Period 1 - CTP-543 12 mg BID: Participants received CTP-543 12 mg tablets, orally, BID, for up to 24 weeks.
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID
Number analyzed (Participants) | 178 | 135
Percentage of participants
  Week 12 | 24.0 [17.6 to 30.4] | 40.2 [31.6 to 48.7]
  Week 16 | 26.9 [20.2 to 33.7] | 39.1 [30.6 to 47.5]
  Week 20 | 25.6 [18.9 to 32.3] | 52.0 [43.2 to 60.9]
  Week 24 | 28.8 [21.9 to 35.8] | 48.7 [39.8 to 57.7]
Statistical Analysis 1: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 12; Test type: Superiority; Difference in percentages = 16.2, 95% CI 2-sided [5.5 to 26.8] — Treatment difference is calculated as the difference between the percentage of responders in the 12 mg BID group versus the 8 mg BID group
Statistical Analysis 2: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 16; Test type: Superiority; Difference in percentages = 12.1, 95% CI 2-sided [1.3 to 22.9] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 20; Test type: Superiority; Difference in percentages = 26.4, 95% CI 2-sided [15.4 to 37.5] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 24; Test type: Superiority; Difference in percentages = 19.9, 95% CI 2-sided [8.5 to 31.3] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Part A, Period 1: Percentage of Participants Who Achieved an Absolute SALT Score ≤20 at Weeks 4, 8, 12, 16, 20, and 24
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: Efficacy population included all participants who were randomized in the study and dispensed study drug during the treatment period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID
Number analyzed (Participants) | 178 | 135
Percentage of participants
  Week 4 | 0 [NA to NA] — Not estimable as 0 participants achieved SALT score criteria of ≤20 | 0 [NA to NA] — Not estimable as 0 participants achieved SALT score criteria of ≤20
  Week 8 | 1.7 [0.0 to 3.7] | 2.3 [0.0 to 5.0]
  Week 12 | 5.8 [2.3 to 9.3] | 16.4 [10.0 to 22.8]
  Week 16 | 10.2 [5.6 to 14.8] | 24.2 [16.8 to 31.6]
  Week 20 | 15.9 [10.3 to 21.4] | 35.2 [26.8 to 43.7]
  Week 24 | 22.1 [15.7 to 28.5] | 42.9 [34.0 to 51.7]
Statistical Analysis 1: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 8; Test type: Superiority; Difference in percentages = 0.6, 95% CI 2-sided [-2.7 to 3.9] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 12; Test type: Superiority; Difference in percentages = 10.6, 95% CI 2-sided [3.3 to 17.9] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 16; Test type: Superiority; Difference in percentages = 14.0, 95% CI 2-sided [5.3 to 22.8] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 20; Test type: Superiority; Difference in percentages = 19.4, 95% CI 2-sided [9.2 to 29.5] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 24; Test type: Superiority; Difference in percentages = 20.8, 95% CI 2-sided [9.8 to 31.7] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Part A, Period 1: Relative Change in SALT Scores From Baseline at Weeks 4, 8, 12, 16, 20, and 24
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss). Relative change (percent change) to baseline is calculated as: 100 x ([post-baseline SALT score - baseline SALT score]/baseline SALT score). Negative change indicates no hair loss.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Efficacy population included all participants who were randomized in the study and dispensed study drug during the treatment period. Overall number of participants analyzed indicates the number of participants with data available for analysis of this outcome measure. Number analyzed indicates the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID
Number analyzed (Participants) | 177 | 132
Percent change
  Relative Change From Baseline at Week 4 | -0.5 (11.17) | -1.0 (8.73)
  Relative Change From Baseline at Week 8: number analyzed (Participants) | 173 | 128
  Relative Change From Baseline at Week 8 | -7.4 (18.41) | -14.8 (21.67)
  Relative Change From Baseline at Week 12: number analyzed (Participants) | 172 | 128
  Relative Change From Baseline at Week 12 | -18.1 (27.42) | -30.9 (33.69)
  Relative Change From Baseline at Week 16: number analyzed (Participants) | 167 | 128
  Relative Change From Baseline at Week 16 | -26.3 (31.68) | -39.9 (36.24)
  Relative Change From Baseline at Week 20: number analyzed (Participants) | 164 | 122
  Relative Change From Baseline at Week 20 | -32.1 (34.26) | -49.0 (37.44)
  Relative Change From Baseline at Week 24: number analyzed (Participants) | 163 | 119
  Relative Change From Baseline at Week 24 | -38.2 (36.85) | -55.3 (38.01)
Statistical Analysis 1: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 4; Test type: Superiority; Least Square (LS) Mean Difference = -0.5, 95% CI 2-sided [-2.8 to 1.8], Standard Error of Mean 1.18 — LS means,standard error(SE),and confidence intervals(CIs) are based on mixed model repeated measures(MMRM)analysis with effects for treatment,visit,treatment-by-visit interaction,and baseline value.The Model uses an unstructured covariance structure
Statistical Analysis 2: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 8; Test type: Superiority; LS Mean Difference = -7.3, 95% CI 2-sided [-11.9 to -2.7], Standard Error of Mean 2.32 — LS means, SE, and CIs are based on an MMRM analysis with effects for treatment, visit, treatment-by-visit interaction, and baseline value. The model is fit using an unstructured covariance structure
Statistical Analysis 3: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 12; Test type: Superiority; LS Mean Difference = -12.4, 95% CI 2-sided [-19.3 to -5.5], Standard Error of Mean 3.50 — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 4: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 16; Test type: Superiority; LS Mean Difference = -14.6, 95% CI 2-sided [-22.2 to -6.9], Standard Error of Mean 3.90 — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 5: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 20; Test type: Superiority; LS Mean Difference = -15.4, 95% CI 2-sided [-23.7 to -7.2], Standard Error of Mean 4.20 — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 6: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 24; Test type: Superiority; LS Mean Difference = -15.4, 95% CI 2-sided [-24.0 to -6.8], Standard Error of Mean 4.36 — [estimate comment as in outcome 8, analysis 2]

9. Secondary Outcome: Part A, Period 1: Percentage of Responders Assessed Using the Clinician Global Impression of Improvement (CGI-I) at Weeks 12, 16, 20 and 24
Description: The CGI-I is a questionnaire that asks the clinician to evaluate the improvement or worsening of the participant's alopecia areata as compared to the start of the study on a 7-point scale. Responses range from 1 (very much worse) to 7 (very much improved). Responders were defined as participants with responses of 6 (much improved) or 7 (very much improved).
Time Frame: Weeks 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID
Number analyzed (Participants) | 178 | 135
Percentage of responders
  Week 12 | 26.7 [20.1 to 33.4] | 47.6 [38.9 to 56.3]
  Week 16 | 37.7 [30.4 to 45.1] | 51.6 [42.9 to 60.2]
  Week 20 | 47.6 [39.2 to 55.2] | 63.1 [54.6 to 71.7]
  Week 24 | 50.3 [42.6 to 58.0] | 64.7 [56.1 to 73.3]
Statistical Analysis 1: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 12; Test type: Superiority; Difference in percentages = 20.9, 95% CI 2-sided [9.9 to 31.8] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 16; Test type: Superiority; Difference in percentages = 13.8, 95% CI 2-sided [2.5 to 25.2] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 20; Test type: Superiority; Difference in percentages = 15.6, 95% CI 2-sided [4.1 to 27.0] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 24; Test type: Superiority; Difference in percentages = 14.4, 95% CI 2-sided [2.9 to 25.9] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: Part A, Period 1: Percentage of Responders Assessed Using the Patient Global Impression of Improvement (PGI-I) at Weeks 12, 16, 20, and 24
Description: The PGI-I is a self-administered questionnaire that asks the participant to evaluate the improvement or worsening of their alopecia areata as compared to the start of the study on a 7-point scale. Responses range from 1 (very much worse) to 7 (very much improved). Responders were defined as participants with responses of 6 (much improved) or 7 (very much improved). PGI responder is a response of 'very much improved' or 'much improved'.
Time Frame: Weeks 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID
Number analyzed (Participants) | 178 | 135
Percentage of responders
  Week 12 | 29.8 [23.0 to 36.7] | 52.8 [44.1 to 61.4]
  Week 16 | 33.5 [26.4 to 40.7] | 55.5 [46.9 to 64.1]
  Week 20 | 40.9 [33.3 to 48.4] | 63.4 [54.9 to 71.9]
  Week 24 | 46.0 [38.4 to 53.7] | 65.5 [57.0 to 74.1]
Statistical Analysis 1: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 12; Test type: Superiority; Difference in percentages = 22.9, 95% CI 2-sided [11.9 to 34.0] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 16; Test type: Superiority; Difference in percentages = 21.9, 95% CI 2-sided [10.7 to 33.1] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 20; Test type: Superiority; Difference in percentages = 22.6, 95% CI 2-sided [11.2 to 33.9] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 24; Test type: Superiority; Difference in percentages = 19.5, 95% CI 2-sided [8.1 to 31.0] — [estimate comment as in outcome 6, analysis 1]

11. Secondary Outcome: Part A, Period 1: Change in the Clinician Global Impression of Severity (CGI-S) Scores From Baseline at Weeks 12, 16, 20, and 24
Description: The CGI-S is a questionnaire that asks the clinician to evaluate the symptom severity of the participant's alopecia areata at the time of assessment. The symptom severity was rated on a scale ranging from 1 to 7, where 1=normal, no hair loss; 2=borderline hair loss; 3=mild hair loss; 4=moderate hair loss; 5=marked hair loss; 6=severe hair loss; 7=among the most extreme hair loss. Higher scores indicate more hair loss. A negative change from baseline indicates less hair loss.
Time Frame: Baseline, Weeks 12, 16, 20, and 24
Population: Efficacy population included all participants who were randomized, dispensed study drug, and had at least 1 post-treatment SALT assessment. Overall number of participants analyzed indicates the number of participants with data available for analysis of this outcome measure. Number analyzed indicates the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID
Number analyzed (Participants) | 172 | 130
Score on a scale
  Baseline | 6.4 (0.78) | 6.3 (0.95)
  Change From Baseline at Week 12: number analyzed (Participants) | 172 | 127
  Change From Baseline at Week 12 | -0.8 (1.15) | -1.4 (1.63)
  Change From Baseline at Week 16: number analyzed (Participants) | 167 | 128
  Change From Baseline at Week 16 | -1.1 (1.37) | -1.8 (1.74)
  Change From Baseline at Week 20: number analyzed (Participants) | 164 | 122
  Change From Baseline at Week 20 | -1.3 (1.38) | -2.1 (1.84)
  Change From Baseline at Week 24: number analyzed (Participants) | 163 | 119
  Change From Baseline at Week 24 | -1.6 (1.64) | -2.4 (1.92)
Statistical Analysis 1: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 12; Test type: Superiority; LS Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.3], Standard Error of Mean 0.16 — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 2: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 16; Test type: Superiority; LS Mean Difference = -0.7, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.18 — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 20; Test type: Superiority; LS Mean Difference = -0.8, 95% CI 2-sided [-1.2 to -0.4], Standard Error of Mean 0.19 — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 4: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 24; Test type: Superiority; LS Mean Difference = -0.7, 95% CI 2-sided [-1.2 to -0.3], Standard Error of Mean 0.20 — [estimate comment as in outcome 8, analysis 2]

12. Secondary Outcome: Part A, Period 1: Change in the Patient Global Impression of Severity (PGI-S) Scores From Baseline at Weeks 12, 16, 20, and 24
Description: The PGI-S is a self-administered questionnaire that asks the participant to evaluate the symptom severity of their alopecia areata at the time of assessment. Symptom severity was rated on a scale ranging from 1 to 7, where 1=normal, no hair loss; 2=borderline hair loss; 3=mild hair loss; 4=moderate hair loss; 5=marked hair loss; 6=severe hair loss; 7=among the most extreme hair loss. Higher scores indicate more hair loss. A negative change from baseline indicates less hair loss.
Time Frame: Baseline, Weeks 12, 16, 20, and 24
Population: The Efficacy Population included all participants who were randomized, dispensed study drug, and had at least 1 post-treatment SALT assessment. Overall number of participants analyzed indicates the number of participants with data available for analysis of this outcome measure. Number analyzed indicates the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID
Number analyzed (Participants) | 172 | 130
Score on a scale
  Baseline | 6.4 (0.75) | 6.4 (0.84)
  Change From Baseline at Week 12: number analyzed (Participants) | 171 | 127
  Change From Baseline at Week 12 | -0.8 (1.31) | -1.1 (1.56)
  Change From Baseline at Week 16: number analyzed (Participants) | 167 | 128
  Change From Baseline at Week 16 | -1.0 (1.41) | -1.6 (1.74)
  Change From Baseline at Week 20: number analyzed (Participants) | 164 | 123
  Change From Baseline at Week 20 | -1.1 (1.41) | -2.1 (1.78)
  Change From Baseline at Week 24: number analyzed (Participants) | 163 | 119
  Change From Baseline at Week 24 | -1.4 (1.66) | -2.3 (1.95)
Statistical Analysis 1: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 12; Test type: Superiority; Least Square (LS) Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.16 — LS means, SE, and CIs are based on an MMRM analysis with effects for treatment, visit, treatment-by-visit interaction, baseline value, and baseline SALT score. The model is fit using an unstructured covariance structure
Statistical Analysis 2: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 16; Test type: Superiority; LS Mean Difference = -0.7, 95% CI 2-sided [-1.0 to -0.3], Standard Error of Mean 0.18 — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 20; Test type: Superiority; LS Mean Difference = -0.8, 95% CI 2-sided [-1.2 to -0.5], Standard Error of Mean 0.18 — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Week 24; Test type: Superiority; LS Mean Difference = -0.8, 95% CI 2-sided [-1.2 to -0.4], Standard Error of Mean 0.21 — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Part A, Period 1: Change in the Individual Items of the Hair Quality Patient Reported Outcome (QPRO) Scale From Baseline at Weeks 12, 16, 20, and 24
Description: The QPRO questionnaire provides additional details on key attributes of hair and helps provide context to the SPRO response. The individual items of QPRO are: Satisfied thickness hair coverage; Satisfied evenness hair coverage; How satisfied with your eyebrows; How satisfied with your eyelashes, scored on a scale ranging from 1 to 5 where 1=very satisfied, 2=satisfied, 3=neither satisfied nor dissatisfied, 4=dissatisfied, 5=very dissatisfied. Higher scores indicates the greater dissatisfaction on hair quality. A negative change from baseline indicate the greater satisfaction on hair quality.
Time Frame: Baseline, Weeks 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID
Number analyzed (Participants) | 172 | 130
Score on a scale
  Satisfied Thickness Hair Coverage: Baseline | 4.6 (0.74) | 4.6 (0.67)
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 12: number analyzed (Participants) | 171 | 127
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 12 | -0.9 (1.17) | -1.3 (1.15)
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 16: number analyzed (Participants) | 167 | 128
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 16 | -1.0 (1.15) | -1.5 (1.14)
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 20: number analyzed (Participants) | 164 | 123
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 20 | -1.1 (1.23) | -1.7 (1.16)
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 24: number analyzed (Participants) | 163 | 119
  Satisfied Thickness Hair Coverage: Change From Baseline at Week 24 | -1.2 (1.38) | -1.7 (1.25)
  Satisfied Evenness Hair Coverage: Baseline | 4.7 (0.62) | 4.7 (0.64)
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 12: number analyzed (Participants) | 171 | 127
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 12 | -0.8 (1.09) | -1.3 (1.09)
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 16: number analyzed (Participants) | 167 | 128
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 16 | -0.9 (1.07) | -1.4 (1.14)
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 20: number analyzed (Participants) | 164 | 123
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 20 | -1.0 (1.11) | -1.6 (1.19)
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 24: number analyzed (Participants) | 163 | 119
  Satisfied Evenness Hair Coverage: Change From Baseline at Week 24 | -1.1 (1.22) | -1.7 (1.18)
  How Satisfied With Your Eyebrows: Baseline | 4.0 (1.23) | 4.1 (1.35)
  How Satisfied With Your Eyebrows: Change From Baseline at Week 12: number analyzed (Participants) | 171 | 127
  How Satisfied With Your Eyebrows: Change From Baseline at Week 12 | -0.8 (1.20) | -1.4 (1.43)
  How Satisfied With Your Eyebrows: Change From Baseline at Week 16: number analyzed (Participants) | 167 | 128
  How Satisfied With Your Eyebrows: Change From Baseline at Week 16 | -1.0 (1.17) | -1.4 (1.44)
  How Satisfied With Your Eyebrows: Change From Baseline at Week 20: number analyzed (Participants) | 164 | 123
  How Satisfied With Your Eyebrows: Change From Baseline at Week 20 | -1.0 (1.28) | -1.5 (1.32)
  How Satisfied With Your Eyebrows: Change From Baseline at Week 24: number analyzed (Participants) | 163 | 119
  How Satisfied With Your Eyebrows: Change From Baseline at Week 24 | -1.1 (1.29) | -1.7 (1.42)
  How Satisfied With Your Eyelashes: Baseline | 3.7 (1.40) | 3.7 (1.44)
  How Satisfied With Your Eyelashes: Change From Baseline at Week 12: number analyzed (Participants) | 171 | 127
  How Satisfied With Your Eyelashes: Change From Baseline at Week 12 | -0.7 (1.12) | -1.1 (1.42)
  How Satisfied With Your Eyelashes: Change From Baseline at Week 16: number analyzed (Participants) | 167 | 128
  How Satisfied With Your Eyelashes: Change From Baseline at Week 16 | -0.8 (1.25) | -1.3 (1.42)
  How Satisfied With Your Eyelashes: Change From Baseline at Week 20: number analyzed (Participants) | 164 | 123
  How Satisfied With Your Eyelashes: Change From Baseline at Week 20 | -0.8 (1.22) | -1.4 (1.37)
  How Satisfied With Your Eyelashes: Change From Baseline at Week 24: number analyzed (Participants) | 163 | 119
  How Satisfied With Your Eyelashes: Change From Baseline at Week 24 | -0.9 (1.28) | -1.5 (1.41)
Statistical Analysis 1: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Satisfied Thickness Hair Coverage: Week 12; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.13 — LS means, SEs, and CIs are based on a mixed model repeated measures analysis with effects for treatment, visit, treatment-by-visit interaction, baseline value, and baseline SALT score. The model is fit using an unstructured covariance structure
Statistical Analysis 2: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Satisfied Thickness Hair Coverage: Week 16; Test type: Superiority; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.13 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Satisfied Thickness Hair Coverage: Week 20; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.3], Standard Error of Mean 0.13 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Satisfied Thickness Hair Coverage: Week 24; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.14 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Satisfied Evenness Hair Coverage: Week 12; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.3], Standard Error of Mean 0.12 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Satisfied Evenness Hair Coverage: Week 16; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.3], Standard Error of Mean 0.12 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Satisfied Evenness Hair Coverage: Week 20; Test type: Superiority; LS Mean Difference = -0.6, 95% CI 2-sided [-0.8 to -0.3], Standard Error of Mean 0.13 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; Satisfied Evenness Hair Coverage: Week 24; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.3], Standard Error of Mean 0.14 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 9: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; How Satisfied With Your Eyebrows: Week 12; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.14 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 10: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; How Satisfied With Your Eyebrows: Week 16; Test type: Superiority; LS Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.13 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 11: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; How Satisfied With Your Eyebrows: Week 20; Test type: Superiority; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.14 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 12: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; How Satisfied With Your Eyebrows: Week 24; Test type: Superiority; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.14 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 13: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; How Satisfied With Your Eyelashes: Week 12; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.13 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 14: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; How Satisfied With Your Eyelashes: Week 16; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.13 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 15: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; How Satisfied With Your Eyelashes: Week 20; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.13 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 16: Comparison: Part A: Period 1 - CTP-543 8 mg BID vs Part A: Period 1 - CTP-543 12 mg BID; How Satisfied With Your Eyelashes: Week 24; Test type: Superiority; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.3], Standard Error of Mean 0.14 — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Part B: Percentage of Participants Who Achieved Restoration of Regrowth Criteria at Weeks 4, 8, 12, 16, 20, and 24
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss). ROR is defined as the participant's attainment of an absolute SALT score of ≤20 during re-treatment.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24 of re-treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part B: CTP-543 8 mg to 4 mg BID to 8 mg BID: Participants who received CTP-543 8 mg during Period 1, followed by CTP-543 4 mg during Period 2 of Part A and met the criteria for loss of regrowth maintenance (LOM) (absolute SALT score of > 20), received re-treatment with CTP-543 8 mg tablets, orally, BID, for up to 24 weeks.
Arm/Group | Part B: CTP-543 8 mg to 4 mg BID to 8 mg BID | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID
Number analyzed (Participants) | 5 | 8 | 15 | 19
Percentage of participants
  Week 4 | 60.0 [17.1 to 100.0] | 62.5 [29.0 to 96.0] | 26.7 [4.3 to 49.0] | 15.8 [0.0 to 32.2]
  Week 8 | 100.0 [100.0 to 100.0] | 62.5 [29.0 to 96.0] | 23.1 [0.2 to 46.0] | 16.7 [0.0 to 33.9]
  Week 12 | 80.0 [44.9 to 100.0] | 62.5 [29.0 to 96.0] | 30.8 [5.7 to 55.9] | 43.8 [19.4 to 68.1]
  Week 16 | 60.0 [17.1 to 100.0] | 62.5 [29.0 to 96.0] | 50.0 [21.7 to 78.3] | 61.1 [38.6 to 83.6]
  Week 20 | 60.0 [17.1 to 100.0] | 62.5 [29.0 to 96.0] | 69.2 [44.1 to 94.3] | 70.6 [48.9 to 92.2]
  Week 24 | 60.0 [17.1 to 100.0] | 50.0 [15.4 to 84.6] | 76.9 [54.0 to 99.8] | 77.8 [58.6 to 97.0]

15. Secondary Outcome: Part B: Relative Change in SALT Scores From Part B Baseline at Weeks 4, 8, 12, 16, 20, and 24
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss). Relative change (percent change) to baseline is calculated as: 100 x ([post-baseline SALT score - baseline SALT score]/baseline SALT score).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24 of re-treatment
Population: Efficacy Population included all participants who were randomized, dispensed study drug, and had at least 1 post-treatment SALT assessment. Number analyzed indicates the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID
Number analyzed (Participants) | 5 | 8 | 15 | 19
Percent change
  Relative Change From Baseline at Week 4 | -20.8 (15.27) | -1.5 (69.43) | 12.1 (39.44) | 47.8 (71.19)
  Relative Change From Baseline at Week 8: number analyzed (Participants) | 5 | 8 | 13 | 18
  Relative Change From Baseline at Week 8 | -39.6 (20.33) | 26.2 (109.97) | 10.5 (48.10) | 47.1 (94.35)
  Relative Change From Baseline at Week 12: number analyzed (Participants) | 5 | 8 | 13 | 16
  Relative Change From Baseline at Week 12 | -42.6 (27.06) | -2.6 (78.81) | -7.2 (84.41) | 33.9 (119.41)
  Relative Change From Baseline at Week 16: number analyzed (Participants) | 5 | 8 | 12 | 18
  Relative Change From Baseline at Week 16 | -48.8 (52.66) | -11.4 (78.88) | -13.4 (95.31) | -15.2 (116.20)
  Relative Change From Baseline at Week 20: number analyzed (Participants) | 5 | 8 | 13 | 17
  Relative Change From Baseline at Week 20 | -54.8 (43.90) | -7.8 (83.35) | -29.2 (93.24) | -31.5 (108.97)
  Relative Change From Baseline at Week 24: number analyzed (Participants) | 5 | 8 | 13 | 18
  Relative Change From Baseline at Week 24 | -39.3 (53.48) | -7.9 (81.41) | -39.3 (84.49) | -38.4 (105.80)

16. Secondary Outcome: Number of Participants Experiencing at Least One Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the patient's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an adverse event. TEAEs were defined as any adverse event that occurs after administration of the first dose of study drug in each Part/Period (ie, on or after the day of the first dose in each Part/Period). TEAEs included both serious and non-serious TEAEs.
Time Frame: From first dose of study drug up to last follow up visit (Week 76)
Population: Safety population included all participants who received study drug during the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID | Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID | Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID | Part A: Period 2 - CTP-543 8 mg BID to Placebo | Part A: Period 2 - CTP-543 12 mg BID to Placebo | Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID
Number analyzed (Participants) | 180 | 137 | 18 | 25 | 18 | 25 | 5 | 8 | 15 | 19
Participants | 124 | 100 | 9 | 12 | 7 | 11 | 2 | 5 | 12 | 14

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to last follow up visit (Week 76)
Description: All-cause mortality: All randomized participants included all participants who were randomized in the study.
  Adverse events: Safety population included all participants who received study drug during the treatment period.
Groups:
- Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID: Participants who received CTP-543 8 mg during Period 1, followed by CTP-543 4 mg during Period 2 of Part A and met the criteria for loss of regrowth maintenance (LOM) (absolute SALT score of > 20), received re-treatment with CTP-543 8 mg tablets, orally, BID, for up to 24 weeks.
Arm/Group | Part A: Period 1 - CTP-543 8 mg BID | Part A: Period 1 - CTP-543 12 mg BID | Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID | Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID | Part A: Period 2 - CTP-543 8 mg BID to Placebo | Part A: Period 2 - CTP-543 12 mg BID to Placebo | Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/137 | 0/18 | 0/25 | 0/18 | 0/25 | 0/5 | 0/8 | 0/15 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/180 | 5/137 | 0/18 | 0/25 | 2/18 | 0/25 | 0/5 | 0/8 | 0/15 | 0/19
Other Adverse Events (participants affected / at risk) | 91/180 | 82/137 | 9/18 | 10/25 | 7/18 | 9/25 | 2/5 | 5/8 | 12/15 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Period 1 - CTP-543 8 mg BID (N=180) | Part A: Period 1 - CTP-543 12 mg BID (N=137) | Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID (N=18) | Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID (N=25) | Part A: Period 2 - CTP-543 8 mg BID to Placebo (N=18) | Part A: Period 2 - CTP-543 12 mg BID to Placebo (N=25) | Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID (N=5) | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID (N=8) | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID (N=15) | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID (N=19)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T Wave Inversion (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Period 1 - CTP-543 8 mg BID (N=180) | Part A: Period 1 - CTP-543 12 mg BID (N=137) | Part A: Period 2 - CTP-543 8 mg BID to 4 mg BID (N=18) | Part A: Period 2 - CTP-543 12 mg BID to 8 mg BID (N=25) | Part A: Period 2 - CTP-543 8 mg BID to Placebo (N=18) | Part A: Period 2 - CTP-543 12 mg BID to Placebo (N=25) | Part B: CTP-543 8 mg BID to 4 mg BID to 8 mg BID (N=5) | Part B: CTP-543 12 mg BID to 8 mg BID to 12 mg BID (N=8) | Part B: CTP-543 8 mg BID to Placebo to 8 mg BID (N=15) | Part B: CTP-543 12 mg BID to Placebo to 12 mg BID (N=19)
Asymptomatic COVID-19 (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 23 | 21 | 3 | 5 | 0 | 0 | 0 | 1 | 4 | 4
Folliculitis (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 11 | 10 | 0 | 3 | 0 | 3 | 0 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 3 | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 23 | 17 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 19 | 20 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neutrophil percentage decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 8 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wants to publish study data or results, the publication or presentation must be provided to Concert for review at least 60 days in advance. If Concert needs to file a patent application prior to publication, the publication can be delayed up to 90 days from Sponsor providing notice to the investigator of such need.

DOCUMENTS (2):
  • Study Protocol (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT04784533/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT04784533/SAP_001.pdf